CLINICAL TRIAL: NCT02188277
Title: Multi-center Open Comparative Randomized Trial of Clinical and Neurophysiological Efficacy and Safety of Xeomin (Botulinum Toxin Type A) vs. Botox (Complex of Botulinum Toxin Type A and Hemagglutinin) in Children With Spastic Equine and Equinovarus Foot Deformation in Pediatric Cerebral Palsy
Brief Title: Treatment With Xeomin Versus Botox in Children With Spastic Equine and Equinovarus Foot Deformation in Pediatric Cerebral Palsy
Acronym: XEBEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Collaborators: LLC Merz Pharma, Russia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRZ-R-201212_01001_N_2
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Cerebral Palsy; Spastic Paraplegia and Hemiparesis; Equine and Equinovarus Foot Deformation
MeSH Terms: conditions — Cerebral Palsy; Paraplegia; Paresis | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xeomin® (Experimental): 4-8 Units per kg body weight. Single injection cycle.
  Interventions: Drug: Xeomin
- Botox® (Active Comparator): 4-6(8) Units per kg body weight. Single injection cycle.
  Interventions: Drug: Botox®

INTERVENTIONS:
Drug: Xeomin — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Administration route is intramuscular injection into medial (two points) and lateral heads (two points) of gastrocnemius.
  Other Names: IncobotulinumtoxinA; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: Xeomin®
Drug: Botox® — Administration route is intramuscular injection into medial (two points) and lateral heads (two points) of gastrocnemius.
  Other Names: OnabotulinumtoxinA
  Arms: Botox®

SUMMARY:
1. To assess the clinical and neurophysiological efficacy of Xeomin® vs. Botox® in children with spastic equine and equinovarus foot deformation in pediatric cerebral palsy
2. To assess the safety of Xeomin® use as compared to Botox® in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 through 12 years of age, of both sexes, suffering from spastic paraplegia or hemiparesis in pediatric cerebral palsy.
* Equine and equinovarus foot posture.
* Gastrocnemius spasticity of 2 points and greater, by modified Ashworth scale.
* Patient can walk unassisted or with a support.
* Mental development of patients is normal or mildly retarded.
* Previous course of spasticity treatment with BTA products was completed earlier than at 6 months before this trial or never administered before.
* Patient's parents have signed an informed consent, are able and wishing to adhere to procedures described in the trial protocol and to the schedule of visits throughout the entire period of treatment.

Exclusion Criteria:

* Fixed ankle joint contracture.
* Previous denervation of spastic muscles by surgery, phenol or alcohol;
* Athetosis and dystonia in the area of injected muscles.
* Inflammation at the planned injection site.
* Elevated body temperature and acute (infectious and non-infectious) diseases at the time of injection.
* Neuromuscular transmission disorders (myasthenia gravis, Lambert-Eaton syndrome, etc.).
* Decompensated physical diseases potentially affecting the trial findings.
* Acute fever, infection or surgery within 1 month before the trial.
* Use of aminoglycosides or spectinomycin within 1 month before starting the trial.
* Hypersensitivity to any of product ingredients.
* Positive history for allergies (especially with regard to protein-containing products).
* Patient's parents are unable or unwilling to adhere to the trial protocol requirements including signing the informed consent and conforming to the schedule of visits.
* Participation in other clinical trials in the last 4 weeks before inclusion.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the degree of spasticity in gastrocnemius according to modified Ashworth scale (AS) | From baseline to day 30
  The AS is a well known and commonly used scale in clinical trials with spasticity. In spastic muscles the resistance to passive movement is assessed. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).

SECONDARY OUTCOMES:
Changes from baseline in patient percentage in groups by the degree of gastrocnemius spasticity according to modified Ashworth scale | From baseline up to day 90
Percentage of decrease in M-response magnitude and area recorded from the lateral and medial gastrocnemius heads, from baseline values | From baseline up to day 90
  Electromyography: The amplitude of a compound muscle action potential (M-wave) is recorded. An electrical stimulation is considered supramaximal when the M-wave amplitude no longer increases while increasing the stimulus. The measurements include the M-wave amplitude and the negative peak area of the M-wave.
Changes from baseline in the ratio of M-response recorded from the lateral and medial gastrocnemius heads and from tibialis anterior | From baseline up to day 90
Changes from baseline in angles and angle ratio of ankle joints at passive and voluntary extension | From baseline up to day 90
Changes from baseline in motor activity according to Gross Motor Function Classification Systems (GMFCS) criteria | From baseline up to day 90
  GMFCS is a 5-level classification system that is a standardized observational instrument for children with CP developed to measure change in gross motor function over time.
Changes from baseline in the degree of spasticity in gastrocnemius according to modified Ashworth scale | Baseline up to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — LLC Merz Pharma, Russia
Locations (3):
- Russia (3):
  - State Budget Institution of Health in Moscow "Scientific and Practical Center of Pediatric psychoneurology Moscow Health Department", Moscow
  - Federal State Autonomous Institution "Scientific Center of Children's Health" of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Budget Educational Institution of Higher Professional Learning "Stavropol State Medical University" of the Ministry of Health of the Russian Federation, Stavropol